CLINICAL TRIAL: NCT06977191
Title: The Role of Perioperative Heart Rate Variability in Predicting Rebound Pain After Total Knee Arthroplasty: A Prospective Observational Study
Brief Title: Heart Rate Variability as a Predictor of Rebound Pain Following Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Mahmut Sami TUTAR, Associate Professor, Department of Anesthesiology and Reanimation, Konya City Hospital
Other Study IDs: 10.04.2025/ 05-605-03
Record Dates: First submitted 2025-05-07; First posted 2025-05-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Rebound Pain; Total Knee Arthroplasty; Postoperative Pain, Chronic; Heart Rate Variability
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate whether heart rate variability (HRV), a marker of autonomic nervous system activity, can predict the occurrence of rebound pain after total knee arthroplasty (TKA). Rebound pain is defined as a sudden and intense pain episode (NRS ≥7) that typically arises after the resolution of peripheral nerve blocks used for postoperative analgesia.

Patients undergoing elective unilateral TKA under spinal anesthesia with peripheral nerve blocks will be included. HRV will be measured both before and after surgery using a chest-worn heart rate monitor. Pain levels, analgesic consumption, sleep quality, and patient satisfaction will also be recorded. The primary goal is to determine whether perioperative HRV values can serve as a predictive biomarker for rebound pain.

Secondary outcomes include the relationship between HRV and pain intensity, opioid use, sleep quality, and length of hospital stay. The findings may contribute to developing individualized pain management strategies for TKA patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* American Society of Anesthesiologists (ASA) physical status I-III
* Scheduled for elective, unilateral total knee arthroplasty under spinal anesthesia
* Planned use of multimodal analgesia including peripheral nerve blocks
* Ability to provide written informed consent
* Ability to understand and complete pain diaries and questionnaires

Exclusion Criteria:

* Known allergy to local anesthetics
* Contraindications to regional anesthesia
* Contraindications to spinal anesthesia
* ASA physical status IV or higher
* Pregnancy or breastfeeding
* Neurological or psychiatric disorders impairing ability to participate or report outcomes
* Use of anticoagulant therapy or presence of coagulation disorders
* Infection at the proposed injection site
* Emergency (non-elective) surgical procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 70 years scheduled for elective unilateral total knee arthroplasty under spinal anesthesia at a tertiary care hospital. All participants will receive multimodal analgesia including peripheral nerve blocks as part of standard care.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Preoperative LF/HF Ratio as a Predictor of Rebound Pain | Preoperative (before spinal anesthesia) to 48 hours postoperative
  To determine whether the preoperative low frequency to high frequency (LF/HF) ratio of heart rate variability is associated with the development of rebound pain after peripheral nerve block resolution. Patients will be classified based on the presence or absence of rebound pain (defined as a shift from NRS ≤3 to ≥7), and mean LF/HF ratios will be compared. Predictive capacity will be evaluated using logistic regression and ROC analysis.

SECONDARY OUTCOMES:
Association Between HRV Parameters and Pain Intensity | 0-48 hours postoperative
  Correlation between perioperative HRV values (SDNN, RMSSD, LF/HF) and postoperative pain scores (measured by NRS at 8h, 12h, 16h, 24h, and 48h).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Tutar, MD, Principal Investigator — KONYA CITY HOSPİTAL
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared due to institutional policy and patient confidentiality considerations.